CLINICAL TRIAL: NCT03973398
Title: 1.1 English Title of Research Project: Comparing the Efficacy of Ultrasound Guided Quadratus Lumborum Block Anterior Subcostal Versus Posterior Approach in Managing Postoperative Pain in Patients Undergoing Nephrectomy Surger: A Prospective Randomized Controlled Double Blinded Study
Brief Title: Anterior vs. Posterior Quadratus Lumborum Block in Nephrectomy Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sherif Mahmoud Mohammed Bekhet (Other)
Responsible Party: Sponsor-Investigator, Sherif Mahmoud Mohammed Bekhet, Principle investigator, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: QLB in Nephrectomy
Record Dates: First submitted 2019-05-21; First posted 2019-06-04 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Quadratus Lumborum Block

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Quadratus Lumborum Block anterior subcostal (QLa) (Active Comparator): Patients in this group will receive Anterior subcostal Quadratus Lumborum block postoperative with 30 ml of 0.125 bupivacaine.
  Interventions: Procedure: Quadratus Lumborum block
- Quadratus Lumborum Block posterior (QLp) (Active Comparator): Patients in this group will receive Posterior Quadratus Lumborum block postoperative with 30 ml of 0.125 bupivacaine.
  Interventions: Procedure: Quadratus Lumborum block
- Quadratus Lumborum Block anterior subcostal control (QLca) (Placebo Comparator): Patients in this group will receive Anterior subcostal Quadratus Lumborum block postoperative with 30 ml of 0.9% normal saline.
  Interventions: Procedure: Quadratus Lumborum block
- Quadratus Lumborum Block posterior control (QLcp) (Placebo Comparator): Patients in this group will receive Anterior subcostal Quadratus Lumborum block postoperative with 30 ml of 0.9% normal saline.
  Interventions: Procedure: Quadratus Lumborum block

INTERVENTIONS:
Procedure: Quadratus Lumborum block — ultrasound guided Quadratus Lumborum block for postoperative pain

SUMMARY:
* Primary outcome: to compare the efficacy of Anterior subcostal versus Posterior approach in ultrasound guided Quadratus Lumborum Block.
* Secondary outcome: to evaluate the efficacy of Quadratus Lumborum Block in the control of postoperative pain in patients undergoing Nephrectomy surgery, hemodynamics, any complications and patients' satisfaction..

DETAILED DESCRIPTION:
A variant of the ultrasound-guided transversus abdominis plane (TAP) block was first described in an abstract, in which local anesthetic injection occurs at the point where the internal oblique and transversus abdominis muscles taper off and adjoin the lateral border of quadratus lumborum (QL) muscle.

Currently, the QL block is performed as one of the perioperative pain management procedures for all generations (pediatrics, pregnant, and adult) undergoing abdominal surgery.

However, there is large disagreement regarding the best approach for administering the block because of unclear mechanisms responsible for the effects and complicated nomenclature system. Nephrectomy for patients with renal cell carcinoma (RCC) was first described in 1969. Surgical treatment varies with the pathology. Simple nephrectomy is the preferred option for those with non-neoplastic disease (e.g. trauma, non-functioning kidney with chronic infection) with radical nephrectomy being preferred in those with neoplastic disease. Radical nephrectomy implies resection of the whole of Gerota's fascia, including the perinephric fat, lymphatics, and the ipsilateral adrenal gland. Here the investigators are going to compare the Anterior (subcostal) approach to the Posterior approach to determine their level of spread and their value in controlling postoperative pain in patients scheduled for Nephrectomy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Both sex
* Age: 18-60 years.
* ASA I and II
* Elective surgery

Exclusion Criteria:

* Patient's refusal.
* Allergy to local anesthetics.
* Peripheral neuropathy.
* Bleeding diathesis.
* Inflammation or infection over injection site.
* Morbid obesity.
* Patients on previous opioid therapy.
* Psychiatric disorders.
* Emergency surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparing the analgesic effects of Anterior subcostal versus Posterior approach in ultrasound guided Quadratus Lumborum Block by using the Numeric Rating Scale. | baseline
  : to compare the efficacy of Anterior subcostal versus Posterior approach in ultrasound guided Quadratus Lumborum Block by The Numeric rating scale (NRS) both resting and ambulatory which measures pain as felt by the patient every two hours for the first 24 hours then every six hours for the second day. the Numeric rating scale is a scale from 0 to 10 with '0' being lowest pain or no pain and '10' is the worst pain felt.
Comparing the analgesic effects of Anterior subcostal versus Posterior approach in ultrasound guided Quadratus Lumborum Block by using the Revised American Pain Society Patient Outcome Questionnaire. | baseline
  to compare the efficacy of Anterior subcostal versus Posterior approach in ultrasound guided Quadratus Lumborum Block by the Revised American Pain Society Patient Outcome Questionnaire which is a set of questions answered by the patient to evaluate the patient's satisfaction and for quality improvement of pain management in hospitalized patients

SECONDARY OUTCOMES:
using the numeric rating scale to determine the effect of Quadratus Lumborum block in reducing the postoperative pain in patients undergoing nephrectomy surgery | baseline
  to evaluate the efficacy of Quadratus Lumborum Block in the control of postoperative pain in patients undergoing Nephrectomy surgery, hemodynamics, any complications and patients' satisfaction.The Numeric rating scale (NRS) both resting and ambulatory which measures pain as felt by the patient every two hours for the first 24 hours then every six hours for the second day. the Numeric rating scale is a scale from 0 to 10 with '0' being lowest pain or no pain and '10' is the worst pain felt.